CLINICAL TRIAL: NCT06468215
Title: Fertility Sparing Therapy for Patients With Stage IA G2 Endometrial Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Deaprtment of Obstetrics and Gynecology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023G2ECFerSp
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Endometrioid; Fertility Preservation
Keywords: endometrial cancer; fertility-sparing treatment; grade 2
MeSH Terms: conditions — Carcinoma, Endometrioid; Endometrial Neoplasms; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study on Fertility Sparing Therapy in IA Stage G2 Endometrial Cancer Patients (Experimental): Treatment Option 1 is a single-drug regimen, with oral medroxyprogesterone acetate (MPA) 500mg/d or MA 320mg/d.
  Interventions: Drug: Treatment Option 1 is a single-drug regimen, with oral medroxyprogesterone acetate (MPA) 500mg/d or MA 320mg/d.
- The Study on Fertility Sparing Therapy in IA Stage G2 Endometrial Cancer Patients (Experimental): Treatment Option 2 is a combination therapy, consisting of oral MPA 500mg/d/MA 320mg/d combined with the intrauterine insertion of the levonorgestrel intrauterine system (LNG-IUS, Mirena IUD).
  Interventions: Drug: Treatment Option 1 is a single-drug regimen, with oral medroxyprogesterone acetate (MPA) 500mg/d or MA 320mg/d.

INTERVENTIONS:
Drug: Treatment Option 1 is a single-drug regimen, with oral medroxyprogesterone acetate (MPA) 500mg/d or MA 320mg/d. — Compare the efficacy of mono-therapy with progesterone versus combined therapy to determine the best treatment option.
  Other Names: Treatment Option 2 is a combination therapy, consisting of oral MPA 500mg/d/MA 320mg/d combined with the intrauterine insertion of the levonorgestrel intrauterine system (LNG-IUS, Mirena IUD).

SUMMARY:
Endometrial cancer (EC) is a prevalent gynecological cancer with an escalating global incidence and a decreasing age of onset. In the era of precision medicine, there is an increasing emphasis on tailoring treatments to different populations to optimize the positive impact of clinical interventions. Fertility-sparing therapies (FST) are gaining popularity for early-stage, low-grade endometrial cancer due to mounting evidence supporting favorable oncologic and pregnancy outcomes. However, consensus regarding the feasibility of fertility-sparing therapy for similar low-risk grade-2 (G2) endometrioid adenocarcinoma remains elusive. Given the uncertainties surrounding fertility-preserving therapy in patients with moderately differentiated endometrial cancer, this study aims to investigate the optimal regimen of fertility-preserving therapy for patients with IAG2.

DETAILED DESCRIPTION:
This study aims to explore effective treatment options and pregnancy outcomes for G2 EC patients who wish to preserve their fertility. It compares the efficacy of monotherapy with progesterone versus combined therapy to determine the best treatment option.

This study is a multi-center, prospective, randomized controlled trial that collects hospital and outpatient records of uterine endometrioid adenocarcinoma patients who undergo fertility-sparing treatment at 10 units from October 2022. The basic items specified in the study are registered.

Selection criteria: Pathological diagnosis of endometrioid adenocarcinoma G2, MRI or ultrasound confirmed localization of the lesion within the endometrium, FIGO (FIGO, 2009) staging IA, age ≤ 45 years, and those who wish to preserve reproductive function, signed informed consent. Exclusion criteria: Tumor invasion of the muscle layer, FIGO (FIGO, 2009) staging IB or higher, tumor differentiation as G1, G3, or non-endometrioid adenocarcinoma, coexistence of malignant tumors in other sites, contraindications or drug prohibitions for conservative treatment, or judged by the investigator to be unsuitable for childbearing. Exclusion criteria: Violation of the treatment protocol; failure to take medication as prescribed, affecting the judgment of drug efficacy; incomplete data affecting the judgment of efficacy and safety. Withdrawal criteria: Intolerance of the used drugs or the appearance of serious complications, including venous or arterial thromboembolism, liver failure, renal failure, anaphylaxis, uterine perforation, etc.; no response to treatment or disease progression during drug therapy; when the patient requests termination of treatment.

Treatment Plan: The treatment plan was randomly divided into two groups. Group 1 was a single-drug treatment plan, with oral medroxyprogesterone acetate (MPA) 500mg/d or megestrol acetate (MA) 320mg/d; Group 2 was a combined treatment plan, with oral MPA 500mg/d/MA 320mg/d combined with the placement of levonorgestrel intrauterine system (LNG-IUS) in the uterus.

Since the treatment began, each 3-6 months is a course. At the end of each course, an endometrial biopsy is performed under hysteroscopy to conduct tissue pathological examination and evaluate the treatment effect. A vaginal color Doppler ultrasound is performed every month, and a pelvic MRI is re-evaluated as needed. Additionally, a side effect assessment is performed for each course, including weight, vaginal bleeding, breast discomfort, gastrointestinal symptoms, liver and kidney function, and thrombosis.

The efficacy assessment is divided into the following categories: (1) Complete Response (CR), (2) Partial Response (PR), (3) Disease Unresponsive or Stable Disease (NC/SD), (4) Disease Progression (PD), and (5) Relapse.

The main measurement indicator is the time required for the first complete remission. The secondary measurement indicators are the one-year complete remission rate, the two-year disease recurrence rate, the cumulative pregnancy rate, pregnancy duration, pregnancy outcomes, changes in serum indicators, and pathological markers.

ELIGIBILITY:
Inclusion Criteria:

* Endometrioid adenocarcinoma G2, diagnosis by pathological.
* The lesion is limited to the endometrium.
* FIGO (2009) staging is IA.
* Age less than 45.
* Strongly request to preserve fertility.
* Sign informed consent.

Exclusion Criteria:

* The tumor has invaded the muscle layer.
* FIGO (2009) stage IB or higher.
* Endometrioid adenocarcinoma G1, G3, or non-endometrioid cancer
* There are malignant tumors in other systems.
* Have contraindications for conservative treatment or drug use.
* Have been judged by the researcher to be unsuitable for childbearing.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female only
Enrollment: 16 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
The Time Required for Complete Remission for the First Time | 5 years
  The time from the diagnosis of G2 endometrioid carcinoma to the first complete remission after fertility-preserving treatment.（year）

SECONDARY OUTCOMES:
One-year complete remission rate | 5 years
  The percentage of patients who achieved complete remission after one year of fertility preservation treatment.
two-year disease recurrence rate | 5 years
  The probability of recurrence within 2 years for patients who underwent treatment for preserving fertility and achieved complete remission.
cumulative pregnancy rate | 5 years
  The percentage of pregnancies that occurred during the observation period.
pregnancy outcome | 5 years
  The pregnancy outcomes in women who successfully conceived after undergoing fertility-sparing treatment. They can be categorized as: full-term delivery; premature delivery; miscarriage; stillbirth.

IPD SHARING:
Plan to Share IPD: No